CLINICAL TRIAL: NCT07397052
Title: The Effect of Mindfulness-Based Nursing Intervention on Anxiety and Vital Signs in Patients Undergoing Open Heart Surgery: A Randomized Controlled Trial
Brief Title: Mindfulness-Based Nursing Care and Anxiety in Open Heart Surgery Patients
Acronym: OH-MIND
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, FİRDEVS EBRU ÖZDEMİR, PhD, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OPENHEART-MINDFULNESS-2026; Ethics Approval No: 2026/062 (Other: Mersin University Health Sciences Research Ethics Committee)
Record Dates: First submitted 2026-01-29; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Open Heart Surgery; Anxiety
Keywords: Mindfulness; Anxiety; Vital Signs; Nursing Care
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care Control Group (Other): Participants in the control group will receive standard perioperative nursing care routinely provided in the clinic. No additional mindfulness or psycho-educational intervention will be administered. Anxiety levels and vital signs will be assessed at the same time points as in the intervention group.
  Interventions: Other: Standard Care Control Group
- Mindfulness-Based Nursing Intervention Group (Experimental): Participants in the intervention group will receive a three-session mindfulness-based nursing intervention delivered individually by a trained nurse. The first session will be conducted one day before surgery, and the second and third sessions will be conducted on postoperative day 1 and postoperative day 2, respectively, after extubation when the patient is cooperative and clinically stable.
  Each session will last approximately 15-20 minutes and will include guided breathing awareness, relaxation, and body awareness techniques. All sessions will be conducted individually in the patient's room. The intervention is standardized and applied consistently to all participants in the intervention group.
  Interventions: Other: Mindfulness-Based Nursing Intervention Group

INTERVENTIONS:
Other: Mindfulness-Based Nursing Intervention Group — The mindfulness-based nursing intervention consists of three structured individual sessions delivered by a trained nurse. The first session is conducted one day before surgery, and the second and third sessions are conducted on postoperative day 1 and postoperative day 2, respectively, after extubation when the patient is cooperative and hemodynamically stable.
  Each session lasts approximately 15-20 minutes and includes guided breathing awareness, relaxation techniques, and brief body awareness exercises adapted to the perioperative cardiac surgery setting. The intervention focuses on present-moment awareness, non-judgmental attention to bodily sensations, and calming of anxiety-related thoughts.
  All sessions are delivered individually at the patient's bedside in a quiet environment. No prior mindfulness experience is required. The intervention is standardized and applied consistently to all participants in the intervention group.
  Arms: Mindfulness-Based Nursing Intervention Group
Other: Standard Care Control Group — Participants in the control group will receive standard perioperative nursing care routinely provided in the cardiovascular surgery clinic. This includes routine preoperative preparation, postoperative monitoring, pain management, and nursing care according to institutional protocols. No additional mindfulness, relaxation, or psycho-educational intervention will be provided.
  Arms: Standard Care Control Group

SUMMARY:
This randomized controlled trial aims to evaluate the effect of a mindfulness-based nursing intervention on anxiety levels and vital signs in patients undergoing open-heart surgery during the preoperative and early postoperative periods.

DETAILED DESCRIPTION:
Patients undergoing open-heart surgery may experience high levels of anxiety due to the complexity of the surgical procedure, the intensive care environment, pain, invasive interventions, and the perception of a life-threatening condition. Increased perioperative anxiety has been reported to negatively affect vital signs such as blood pressure, heart rate, and respiratory rate, prolong recovery, and reduce patient comfort.

Although pharmacological methods are commonly used to manage anxiety, they may cause adverse effects including sedation, respiratory depression, and hemodynamic instability. Therefore, non-pharmacological nursing interventions are of particular importance in cardiac surgery patients.

Psychosocial and supportive nursing interventions have been shown to reduce anxiety and support physiological stability. In recent years, mindfulness-based interventions have emerged as safe and feasible approaches to reduce stress and anxiety through breath awareness, relaxation, and present-moment techniques. Previous studies in various surgical populations have demonstrated that mindfulness-based interventions can reduce anxiety levels and positively influence certain physiological parameters. However, randomized controlled trials evaluating structured and short-term mindfulness-based nursing interventions during the preoperative and early postoperative periods in open-heart surgery patients are limited.

This study is designed as a quantitative, randomized controlled trial to evaluate the effects of mindfulness-based nursing interventions applied during the preoperative and early postoperative periods on anxiety levels and vital signs in patients undergoing open-heart surgery. The findings are expected to contribute to evidence-based nursing practices and support clinical care processes in the management of anxiety in cardiac surgery patients.

The mindfulness-based nursing intervention consists of brief, structured sessions focusing on breath awareness, relaxation, and present-moment attention, delivered individually by a trained nurse during the preoperative and early postoperative periods.

Outcome assessments, including anxiety questionnaires and vital sign measurements, will be performed by nurses who are not involved in the intervention and are blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Having a planned elective open heart surgery

  * Being able to communicate in Turkish and understand the given instructions
  * Being conscious, cooperative and oriented
  * Having agreed to participate in the research in the preoperative period
  * Being extubated and hemodynamically stable in the postoperative period

Exclusion Criteria:

* Patients with pre-existing serious psychiatric illnesses (e.g., schizophrenia, bipolar disorder)

  * Patients with cognitive impairment or those unable to complete the STAI-S scale
  * Patients with neurological or sensory problems that impair hearing, speech, or communication
  * Patients requiring long-term mechanical ventilation in the postoperative period
  * Patients requiring re-intubation in the postoperative period
  * Patients with hemodynamic instability or those monitored under deep sedation in the intensive care unit
  * Patients who develop serious postoperative complications (e.g., stroke, massive bleeding)
  * Patients who refuse to participate in the study or wish to withdraw from the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
State Anxiety Level (STAI-S) | At baseline (preoperative day), postoperative day 1, and postoperative day 2
  Anxiety level will be assessed using the State Anxiety subscale of the State-Trait Anxiety Inventory (STAI-S), a validated self-report scale consisting of 20 items. Total scores range from 20 to 80, with higher scores indicating higher levels of anxiety.

SECONDARY OUTCOMES:
Blood Pressure | At baseline (preoperative day), postoperative day 1, and postoperative day 2
  Systolic and diastolic blood pressure will be measured using standard non-invasive monitoring methods.

OTHER OUTCOMES:
Heart Rate | At baseline (preoperative day), postoperative day 1, and postoperative day 2
  Heart rate will be recorded as beats per minute using routine clinical monitoring.
Respiratory Rate | At baseline (preoperative day), postoperative day 1, and postoperative day 2
  Respiratory rate will be measured as breaths per minute through routine clinical observation.
Oxygen Saturation (SpO2) | At baseline (preoperative day), postoperative day 1, and postoperative day 2
  Peripheral oxygen saturation (SpO2) will be measured as a percentage (%) using pulse oximetry as part of routine monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Firdevs Ebru Özdemir, PhD, Principal Investigator — Mersin University

REFERENCES:
- [Background] Garland EL, Farb NA, Goldin P, Fredrickson BL. Mindfulness Broadens Awareness and Builds Eudaimonic Meaning: A Process Model of Mindful Positive Emotion Regulation. Psychol Inq. 2015 Oct 1;26(4):293-314. doi: 10.1080/1047840X.2015.1064294. Epub 2015 Nov 24. PMID 27087765